CLINICAL TRIAL: NCT05742165
Title: Time Restricted Eating for Weight Loss Maintenance (TWIST): A Single-Site, Pilot Feasibility and Acceptability Randomized Clinical Trial in Adults With Recent Weight Loss
Brief Title: Time Restricted Eating for Weight Loss Maintenance
Acronym: TWIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-01453; K99HL163474 (NIH)
Record Dates: First submitted 2023-02-15; First posted 2023-02-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Obesity
Keywords: weight loss maintenance; intermittent fasting; time-restricted eating; weight-reduced state
MeSH Terms: conditions — Obesity; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-Restricted Eating - 6 Hours (TRE6) (Experimental): Participants will be instructed to consume all daily food and beverages during their allotted 6-hour time period.
  Interventions: Behavioral: Time Restricted Eating (TRE)
- Time-Restricted Eating - 10 Hours (TRE10) (Experimental): Participants will be instructed to consume all daily food and beverages during their allotted 10-hour time period.
  Interventions: Behavioral: Time Restricted Eating (TRE)

INTERVENTIONS:
Behavioral: Time Restricted Eating (TRE) — TRE involves only consuming food and beverages during a particular consecutive time period - in the case of this study, either 6 hours or 10 hours. Participants will self-select the timing of their first eating occasion of the day, with the provision that their first meal of the day will be consumed within 3 hours of their wake- up time and finished no less than 3 hours prior to bed time. During the fasting period, participants will be encouraged to drink water, and will be permitted to consume zero-calorie beverages. Participants will be instructed to self-monitor all eating occasions using the MyCircadianClock (mCC) smartphone app, which date- and time-stamps all food entries. Participants will also be instructed to self-monitor their body weight daily using a Bluetooth-enabled Renpho scale, which permits remote collection of body weight.

SUMMARY:
The aim of this pilot feasibility and acceptability, randomized clinical trial will be to examine the effects of two-time restricted eating (TRE) interventions on weight loss maintenance (WLM). This study will be conducted in 40 individuals with non-surgical weight loss of ≥5% initial body weight recruited from the NYU Langone Health Weight Management Program and NY-MOVE! Weight Management Clinic at the Manhattan VA. Measurements will occur at baseline, 4 and 12 weeks. Participants will be randomized with equal allocation to 2 groups: (1) TRE6 or (2) TRE10. The TRE6 will restrict their eating window to 6 hours per day and the TRE10 to 10 hours per day.

ELIGIBILITY:
Inclusion Criteria:

* ≥5% non-surgical weight loss from NYULH-WMP and NY-MOVE! Endocrinology Weight Management Clinic in the last 3 months
* BMI between 20.5 - 45 m/kg2
* between the ages 25 to 65 years old
* own a smartphone or willing to use a smartphone if provided for self-monitoring
* Eating window >12 h per day
* <150 mins/wk of physical activity
* log at least 2 meals into the smartphone app on ≥5 days

Exclusion Criteria:

* <25 years or >65 years of age
* Body weight in excess of 400lbs (181.4kg)
* pregnant, trying to get pregnant or breastfeeding
* previous or planned bariatric surgery
* previous or current history of eating disorder
* ongoing participation in another weight-management research study
* continued participation in a weight loss program other than the proposed study
* currently on appetite suppressants
* currently following intermittent fasting or skipping meals
* eating window <11h 59min/day
* perform overnight shift work more than once a week
* work that includes travel across one or more time zones
* currently on anti-obesity medications (AOMs) such as, GLP-1 analogues (exenatide, tirzepatide, semaglutide, liraglutide) and pancreatic lipase inhibitors (Orlistat/Xenical and Alli)
* prescribed medications expected to result in weight loss such as Orlistat, Naltrexone, Bupropion, Lorcaserin, Phentermine, Topiramate, or Liraglutide, and who are unwilling to delay treatment with these medications for the next 3 months
* unable or unwilling to provide informed consent
* unable to participate meaningfully in the intervention (e.g., uncorrected sight and hearing impairment)
* unwilling to accept randomization assignment
* unable to log at least 2 meals into the smartphone app on ≥5 d during the screening period
* have type 1 or other conditions that would preclude restricted eating windows
* have type 2 diabetes with a HbA1c >7.0% on medications except for metformin alone
* narcolepsy
* active cancer
* organ dysfunction
* current steroid use
* daytime sleepiness with the Epworth Sleepiness Scale >10
* severe insomnia with a score ≥15 on the Insomnia Severity Index
* >2.5 kg additional weight loss during run-in phase (weight regain is not an exclusion criteria)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Retention Rate | Up to Week 12
  Percentage of participants who complete all study visits. Measure of feasibility.
Recruitment Rate | Up to Week 12
  Number of individuals who must be approached to enroll one participant in the study. A recruitment funnel will be developed by documenting the total number of eligible patients completing the NYU Langone Health-WMP and NY- MOVE! programs losing ≥5% of their baseline body weight.
TRE Experience Questionnaire (TRE-EQ) Score | Week 12
  Online questionnaire that includes 5-point scaled items (0=strongly disagree, 5=strongly agree) regarding difficulties encountered with hunger and appetite; eating within the assigned window; coordinating the TRE window with work, school and home demands; and accommodating social connections (e.g., behaviors and preferences of fellow diners).
Adherence Rate | Up to Week 12
  Using data from participant-worn ActiGraphs and on eating patterns, a day will be labeled "adherent" if all eating occasions (food or beverage with caloric value) are measured inside (± 30 minutes) their prescribed eating window. Adherence rate will be calculated by dividing the total number of adherent days by the total number of days with a logged eating occasion.

SECONDARY OUTCOMES:
Change from Baseline in Lean Mass | Baseline, Week 12
  Measured using Bioelectrical Impedance Analysis (BIA). Expressed in kilograms.
Change from Baseline in Fat Mass | Baseline, Week 12
  Measured using BIA. Expressed in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Mary A. Sevick, ScD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [collin.popp@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to collin.popp@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT05742165/ICF_000.pdf